CLINICAL TRIAL: NCT01279083
Title: A Phase I/II Dose Escalation Safety and Efficacy Trial of DE-112 Ophthalmic Solution in Subjects With Primary Open-Angle Glaucoma or Ocular Hypertension
Brief Title: Safety and Efficacy Trial to Treat Open-Angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Santen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 29-001
Record Dates: First submitted 2011-01-14; First posted 2011-01-19 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-12

CONDITIONS: Open-angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Concentration 1 (Experimental)
  Interventions: Drug: DE-112
- Concentration 2 (Experimental)
  Interventions: Drug: DE-112
- Concentration 3 (Experimental)
  Interventions: Drug: DE-112
- Concentration 4 (Experimental)
  Interventions: Drug: DE-112
- Vehicle Solution (Placebo Comparator)
  Interventions: Drug: DE-112 Vehicle Solution
- Timolol Maleate Ophthalmic Solution (Active Comparator)
  Interventions: Drug: Timolol Maleate Solution

INTERVENTIONS:
Drug: DE-112 — Topical ocular solution
  Arms: Concentration 1
Drug: DE-112 — Topical ocular solution
  Arms: Concentration 2
Drug: DE-112 — Topical ocular solution
  Arms: Concentration 3
Drug: DE-112 — Topical ocular solution
  Arms: Concentration 4
Drug: DE-112 Vehicle Solution — Topical ocular solution
  Arms: Vehicle Solution
Drug: Timolol Maleate Solution — Topical ocular solution
  Arms: Timolol Maleate Ophthalmic Solution

SUMMARY:
To investigate the safety and efficacy of DE-112 in lowering intraocular pressure in subjects with primary open-angle glaucoma or ocular hypertension.

DETAILED DESCRIPTION:
This study will be conducted in two stages. Stage One is an open-label, adaptive dose-selection, safety and efficacy trial of up to four concentrations of DE-112 ophthalmic solution enrolling a total of 24 subjects.

Stage Two of the study is a randomized, double-masked, placebo- and active-controlled, parallel-group, multi-center trial comparing the efficacy and safety of two concentrations of DE-112 ophthalmic solution with placebo and timolol enrolling a total of 120 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Provide signed, written informed consent
* 18 yeas of age and older
* Diagnosed with primary open-angle glaucoma or ocular hypertension
* Female subject of childbearing potential must utilize reliable contraceptive throughout the study and have a negative urine pregnancy test prior to enrollment into this study
* Meet specific Visit 2, Day 0 (Baseline)criteria at baseline

Exclusion Criteria:

* Females who are pregnant, nursing or planning a pregnancy
* Presence of any abnormality or significant illness that could be expected to interfere with the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2011-01; Primary Completion 2011-11 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Intraocular pressure (IOP) | 29 days
  Change from baseline in mean diurnal IOP

SECONDARY OUTCOMES:
Intraocular pressure (IOP) | 29 days
  Percent change from baseline in mean diurnal IOP

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Austin, Texas
  - San Antonio, Texas